CLINICAL TRIAL: NCT04443257
Title: REassessement After Hospitalization for Sars-COV-2 Infection : Standardized Assessment of Sequelae and Comorbidities 3 to 6 Months After Hospitalization
Brief Title: REassessement After Hospitalization for Sars-COV-2 disordER
Acronym: REHCOVER
Status: Terminated | Type: Observational
Why Stopped: not enough inclusions
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0340
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sars-CoV2
Keywords: comorbidities; Sars-CoV2; sequelae; patient outcome assessment; Covid19; quality of life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment of the sequelae after hospitalization for Sars-COV-2 — the incidence of chronic respiratory failure and fibrosis, as well as of comorbidities including cardiovascular, metabolic, renal, hepatic, neurological, and psychological diseases

SUMMARY:
Currently, the sequelae and short-term medical and psychological impact of the sars-cov-2 infection ("CoVID-19") remain poorly described. The clinical and functional sequelae that may persist after acute sars-cov-2 ("CoVID-19") infection are essential to explore, in order to ensure the best possible follow-up of patients after discharge from hospital.

DETAILED DESCRIPTION:
Since sars-cov-2 ("CoVID-19") is a newly defined infection, its sequelae and short-term medical and psychological impact remain poorly described.The clinical and functional sequelae that may persist after acute sars-cov-2 ("CoVID-19") infection are essential to explore, in order to ensure the best possible follow-up of patients after discharge from hospital.

Indeed, some patients may develop chronic respiratory failure, pulmonary fibrosis, or other comorbidities including cardiovascular or metabolic diseases. The psychological impact is also essential to assess. The sequelae and comorbidities of patients could also vary depending on the severity of the initial acute involvement.

Investigators propose to explore the sequelae of patients who have been hospitalized for acute sars-cov-2 infection, between 3 to 6 months after discharge from hospital, by characterizing the incidence of chronic respiratory failure and fibrosis, as well as of various comorbidities such as cardiovascular, metabolic, and psychological diseases.

ELIGIBILITY:
Inclusion Criteria:

* patient who was hospitalized within 3 to 6 months for a sars-CoV infection

Exclusion Criteria:

* Absence of signed informed consent
* pregnancy or breastfeeding
* patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult who was hospitalized within 3 to 6 months for a sars-CoV infection at Montpellier University Hospital
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Development or worsening of a ventilatory disorder and/or chronic respiratory failure assessed by spirometry | 3 to 6 months after Sars coV 2 infection

SECONDARY OUTCOMES:
Assessment of dyspnea | 3 to 6 months after Sars coV 2 infection
  assessed by 0-10 Borg scale
Description of pulmonary lesions as assessed by lung CT scan | 3 to 6 months after Sars coV 2 infection
  assessed by lung CT scan
Development of pulmonary fibrosis as assessed by lung CT scan | 3 to 6 months after Sars coV 2 infection
  assessed by lung CT scan
Incidence or worsening of cardiovascular diseases | 3 to 6 months after Sars coV 2 infection
  assessed by incidence of cardiovascular events, venous thromboembolism, and transthoracic echocardiogram
Incidence or worsening of renal disease | 3 to 6 months after Sars coV 2 infection
  renal function and urinary parameters
Incidence or worsening of liver disease | 3 to 6 months after Sars coV 2 infection
  hepatic blood parameters
Incidence or worsening of psychological pathology : anxiety | 3 to 6 months after Sars coV 2 infection
  assessed by validated scale: Generalized Anxiety Disorder-7 (GAD7)
Incidence or worsening of psychological pathology: depression | 3 to 6 months after Sars coV 2 infection
  assessed by validated scales: Patient Health Questionnaire-9 (PHQ9)
Incidence or worsening of psychological pathology: post-traumatic stress | 3 to 6 months after Sars coV 2 infection
  assessed by validated scale : Post-traumatic Checklist for DSM-5 (PCL-5)
Incidence or worsening of psychological pathology: insomnia | 3 to 6 months after Sars coV 2 infection
  assessed by validated scale : insomnia severity index (ISI)
Assessment of the health-related quality of life | 3 to 6 months after Sars coV 2 infection
  assessed by validated scale (EQ-5D-L questionnaire)
Assessment of the fatigue | 3 to 6 months after Sars coV 2 infection
  assessed by the fatigue severity sale
Assessment of the socioeconomic deprivation | 3 to 6 months after Sars coV 2 infection
  assessed by the Evaluation of Deprivation and Inequalities in Health Examination (EPICES) scale
development or worsening of metabolic disorders: diabetes, thyroid diseases, dyslipidemia, adrenal disorders, malnutrition | 3 to 6 months after Sars coV 2 infection
  assessed by blood glucose level, HbA1C, lipid blood tests, TSH, T3, T4, antithyroperoxydase antibodies, cortisol, ACTH, renin, aldosteron, albumin level, vitamin D level, iron status, weight changes
Development of auto-immune disorders | 3 to 6 months after Sars coV 2 infection
  assessed by lupus anticoagulant, anti-cardiolipin, anti-β2-glycoprotein
Assessment of the evolution of the humoral anti-SARS-CoV-2 immunization profile | 3 to 6 months after Sars coV 2 infection
  Presence and levels of anti-SARS-CoV-2 antibodies of IgG, IgA and IgM isotypes
Patients' self-reported level of physical activity | 3 to 6 months after Sars coV 2 infection
  assessed by the International Physical Activity Questionnaire (IPAQ)
Determination of risk factors associated with sequelae or comorbidities | 3 to 6 months after Sars coV 2 infection

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon a reasonable request
Supporting Information: Study Protocol
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and institutional review board (IRB) review. Dataset will be shared after careful examination by the study board of investigators.

REFERENCES:
- [Result] Berger M, Daubin D, Charriot J, Klouche K, Le Moing V, Morquin D, Halimi L, Jaussent A, Taourel P, Hayot M, Cristol JP, Nagot N, Fesler P, Roubille C. Mid-Term Sequelae of Surviving Patients Hospitalized in Intensive Care Unit for COVID-19 Infection: The REHCOVER Study. J Clin Med. 2023 Jan 28;12(3):1000. doi: 10.3390/jcm12031000. PMID 36769648